CLINICAL TRIAL: NCT04843358
Title: Efficacy of Expressive Writing on Quality of Life Among Breast Cancer Survivors in Oman: A Double Blind Randomized Controlled Trial - A Study Protocol
Brief Title: Efficacy of Expressive Writing on Quality of Life Among Breast Cancer Survivors in Oman: A Double Blind Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Mohammed Al Alawi, Principal Investigator, Dr Mohmmed Al Alawi Bsc, MD, MRCPsych, OMSBPsych, ARABPsych, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14/2021
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Quality of Life; Expressive Writing; Psychological
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Disclosure (Experimental): Participants in the emotional disclosure arm will be told to write continuously for 20 min about their deepest thoughts and feelings regarding their breast cancer experience
  Interventions: Behavioral: Emotional Disclosure
- Non-Emotional Writing (Active Comparator): Participant allocated to the control group will be asked to describe in detail their daily activities in a non-emotional manner in accord with Pennebaker's published instructions
  Interventions: Behavioral: Non-Emotional Writing

INTERVENTIONS:
Behavioral: Emotional Disclosure — The trial member will deliver instructions "For the next three days, I want you to write about your experience with cancer. In your writing, I want you to really let go and explore your very deepest emotions and thoughts. It is critical that you delve deeply. Ideally, I would like you to write about those parts of the experience you found hard to share with others. Perhaps this will provide an opportunity to really examine those thoughts and emotions. You might tie your personal experiences to other parts of your life. How is it related to your family life, relationship with your spouse, your children, your sexuality, daily activities, hobbies, your past, your childhood, your work? These are just some examples."
  Arms: Emotional Disclosure
Behavioral: Non-Emotional Writing — The trial member will deliver instructions were as follows." For the next three days, I want you to write about how you use your time. We are interested in everything you do during the course of a day. In your writing I want you to be completely objective. We are not interested in your emotions or opinions. Feel free to be as detailed as possible
  Arms: Non-Emotional Writing

SUMMARY:
Background Breast cancer is the most common cancer affecting women globally. Additionally, it is the most common cause of cancer mortality among women. Internationally, breast cancer is the most frequently diagnosed cancer among women in 140 of 184 countries. Global registry surveys also demonstrate that the incidence of breast cancer will increase by 46% and affect more than 3,059,829 people by 2040. The rate of breast cancer deaths will increase by 58.3% and affect more than 356,225 women. Psychologically, it has been shown that emotional suppression experienced by some women with breast cancer is highly predictive of low quality of life and psycho-somatic morbidities during the process of treatment. Such attitude towards emotional suppression is thriving well in Arab societies where somatizing, as opposed to psychologizing, distress is prevailing proclivity. Expressive writing may provide a tool to meet such need. Taken together and given the lack of any study exploring EW effect of Quality of life in women with breast cancer. The current study aims to examine the impact of expressive writing on quality of life in a randomized controlled trial among cancer survivor in Oman.

Hypothesis The primary hypothesis states that compared to writing about neutral topic, expressive writing intervention will lead to a better improvement in quality of life among breast cancer patients after two months of the intervention.

Objectives To assess the efficacy of 3 sessions EWI versus Writing about neutral topic, on Quality of life of Breast Cancer Survivors at 1- and 2-month post intervention.

Method This study is a multicenter, prospective, double blind, parallel RCT with a 2-month follow-up and will be carried out at Oman's comprehensive cancer care & research center and Sultan Qaboos University Hospital, Muscat, Oman. Sixty four participants will be randomized to 3 sessions EWI group or neutral topic writing group, using a fixed randomization schedule allocating participant between the two intervention arms in a 1:1 ratio.

DETAILED DESCRIPTION:
Background Breast cancer is the most common cancer affecting women globally. Additionally, it is the most common cause of cancer mortality among women. Internationally, breast cancer is the most frequently diagnosed cancer among women in 140 of 184 countries. Global registry surveys also demonstrate that the incidence of breast cancer will increase by 46% and affect more than 3,059,829 people by 2040. The rate of breast cancer deaths will increase by 58.3% and affect more than 356,225 women.

In the Middle eastern countries, breast cancer is responsible for the highest prevalence rate (21.9%), new incident (17.7%), and mortality (11.6%) caused by different types of neoplasms. In Oman, the incidence rate of breast cancer nearly doubled between 1996 and 2015 from 13.6 to 26.9 per 100 000 women. According to recent data from Ministry of Health, breast cancer is most of common cancer as it accounts for 24.4 percent of all registered cancer incidents in the Sultanate. Such data herald several repercussion at individual and societal levels from health as well as financial dimensions. Health related Quality of life of breast cancer patient is one main concern to be addressed in this context. Health-related quality of life refers to the extent to which one's usual or expected physical, emotional, and social functioning are touched by the cancer or its treatment. The time of diagnosis, initial stages of investigations, the treatment course, and the months following the end of treatment are challenging times for patients both physically and emotionally. During these times, uncertainties, difficulty to adjust and hampered quality of life are inevitable. Women diagnosed with breast cancer are no exception and could endure several emotional and physical challenges. Plethora of literature indicate that the survivorship time, after the surgery undergoing chemotherapy and radiotherapy, is often comes with psychological problems and reduced quality of life (QOL). The reasons for low quality of life among breast cancer population can be conceived of as bio-psycho-social. From biological aspect, chemotherapy side effects play a major a role. These include increased mental and physical symptoms such as anxiety, nausea, constipation, and anemia. Consequently, these side effects can have negative impact of on treatment of breast cancer. Perceived lack of social support, stigma of breast cancer diagnosis, and poor self-image have been recognized as significant moderators of quality of life among breast cancer women.

Psychologically, it has been shown that emotional suppression experienced by some women with breast cancer is highly predictive of low quality of life and psycho-somatic morbidities during the process of treatment. Such attitude towards emotional suppression is thriving well in Arab societies where somatizing, as opposed to psychologizing, distress is prevailing proclivity.

While recognizing the methodological hurdles in discerning and gauging such concepts of emotional suppression , it remains pivotal to delve into interventions to help breast cancer survivors to navigate through these challenges resulting from lengthy process of investigation and treatment. Several psychotherapeutic interventions were tested including Expressive Writing. Expressive Writing is one type of intervention aimed at improving emotion regulation through emotional disclosure. According to the expressive writing intervention (EWI) paradigm, it may be possible to improve both mental and physical health through improving self-regulation of emotion-related experiences.

Many mechanisms have been put forward to explicate the effects of Expressive Writing. Expressive writing may decrease individuals' distress by improving self-regulation of emotions, behaviors, and physiological responses. In some way, expressive writings help the person to connect thoughts to feelings. Furthermore, modulating autonomic arousal to cancer related thoughts and feelings and cognitive processing of events into a coherent and meaningful narrative have been suggested as mechanisms leading to desirable effect of EW. According to the social integration model, expressive writing might encourage individuals to seek social support, which, in turn, feeds in their psychological well-being. In 1986, Pennebaker for the first time used Expressive writing (EW), which a brief emotional disclosure experiment, with college students. st Pennebaker's paradigm for EW experiment encouraged participants to disclose in writing about their trauma-related personally distressing thoughts and feelings for 20 min over four consecutive days and had another group to write about neutral topic. Emotional disclosure arm had shown enhanced well-being and fewer medical visits following writing compared to those who wrote about neutral topics. Pennebaker and Beall (1986) found that EW is a potentially effective intervention which was later tested on various population and settings including, clinically ill patients and healthy individuals. , , .

After Walker's first paper reporting the efficacy of EW with Breast cancer patients, several trials have been launched based Pennebaker's paradigm to provide the unmet needs of this population. , , , In 2006, Frattaroli J et al produced the largest meta-analysis of 146 randomized, controlled trials (RCTs) of different types of experimental disclosure among clinical and healthly populations. The reported an overall effect (r = 0.075≈Cohen's d = 0.15) which was statistically significant. . Ten years later, another review of 20 RCT indicated a significant small effect on improving physical cancer symptoms; however, the effects on psychological and cognitive end points were not significant. However, subgroup analysis showed a significant effect on health-related quality of life between the EW intervention group and the usual care group. Specifically, looking at Breast cancer samples, till the date of writing this background, there have been at least 15 clinical trials and two systematic reviews that explored the rule of expressive writing in alleviating psychological and physical distress among women with breast cancer at different stage of illness. , As with many psychological Interventions, the results of the trials on the efficacy and effectiveness of EW among breast cancer women have not been consistent. The possible reasons are heterogeneous clinical samples, different stages of illness, difference in the Intervention and control conditions, using various outcomes measures, lack of inclusion of a number of mediators including presence/absence of social constraints. Social constraints are the perceived insufficient social assistance resulting in a disinclination to express thoughts and feelings about a specific stressor (e.g., people may respond by minimizing the experience, acting uncomfortable when emotions are expressed, or simply avoiding the person who is attempting to talk about the experience). Given the nature of Arab culture, where social constraints are present13, one could expect that patients with breast cancer may not have avenues to talk about their deep thoughts and feelings in relation to their illness. Therefore, Expressive writing may provide a tool to meet such need. Taken together and given the lack of any study exploring EW effect of Quality of life in women with breast cancer. The current study aims to examine the impact of expressive writing on quality of life in a randomized controlled trial among cancer survivor in Oman. Hypothesis The primary hypothesis states that compared to writing about neutral topic, expressive writing intervention will lead to a better improvement in quality of life among breast cancer patients after two months of the intervention.

Objectives To assess the efficacy of 3 sessions EWI versus Writing about neutral topic, on Quality of life of Breast Cancer Survivors at 1- and 2-month post intervention.

Methods Study Design This study is a multicenter, prospective, double blind, parallel RCT with a 2-month follow-up and will be carried out at Oman's comprehensive cancer care & research center and Sultan Qaboos University Hospital, Muscat, Oman. Participants will be randomized to 3 sessions EWI group or neutral topic writing group, using a fixed randomization schedule allocating participant between the two intervention arms in a 1:1 ratio.

Allocation, concealment, and randomization Block randomization sequence of 6 will be generated using software that will allocate participants in a 1:1 ratio to balance the number of the subjects in each arm. Allocation process will be conducted by centralized service at SQUH with help of independent nurse who is not involve in the research. Participants allocation sequence either in intervention or control arm will be concealed from the study participants and the researchers before the beginning of the trial to avoid selection bias. Each coded sealed opaque envelope which contained participant's treatment allocation will opened by research assistant not involved in the study or the process of data collection or analysis. All participants will have a code number allocated to them. The design of this trial is double blind, the participant will be blinded to the name of the group allocated to. They will be informed that they are participating in writing study for wellbeing in breast cancer women and will be informed that the study aims to capture their inner experiences through writing and will not be made aware of whether they are assigned to an experimental or a control arms. The outcome assessor will be blind to the participant's allocation.

Sample Size The Superiority hypothesis parallel clinical trial model will be adopted to calculate the required sample size in each arm to achieve a mean effect size of d = 0.8, according to published literature, of EWI. Power analysis revealed that 30 participants per group would yield 80% power to test the primary hypothesis with 5% type one error rate. Considering 5% attrition rate, the total needed sample size will be 64.

Eligibility criteria

* Omani Women Having a breast cancer diagnosis stage, I and II
* Completing breast cancer surgery within 5 years
* Subsequently received adjuvant treatment including chemotherapy, hormonal treatment, or Radiation therapy
* Being comfortable writing and speaking in Arabic Exclusion Criteria
* Nonconsenting
* Presence of severe physical illness
* Diagnoses with severe Mental or intellectual disorder
* Advanced case of breast cancer
* Un able to comply with trial protocol
* Presence of another cancer diagnoses

Measure Socio-Demographic Data. This questionnaire contains basic demographic information, including age, marital status, number of children, living with nuclear or extended family, employment, highest education, and presence of financial strain, presence of social support, and presence of social constrain from disclosure.

Medical History Data. Participants will be asked to provide data in relation to their cancer, including date of diagnosis, tumor site, stage of disease at diagnosis, treatments received, and other concurrent chronic health problems and medications. This information will be ascertained through review of patients' medical records Functional Assessment of Cancer Therapy general scale: FACT-G V4 This 27-item measure examines the perceived quality of life across four dimensions including physical, social, emotional, and functional well-being in the past week. The scale was validated among various population of breast cancer survivors globally. Versions of the FACT-G questionnaire are available in 45 different languages, permitting cross-cultural comparisons of people from diverse backgrounds, adopting translation methodology developed for the Functional Assessment of Chronic Illness Therapy (FACIT) project into European, Asian, and African languages (www.facit.org). The internal consistency reliability ranged between 0.71 and 0.82. The test-retest reliability within 24-48 h was found to be 0.80. , The Arabic version was psychometrically tested among Jordanian cancer patients and proved to be valid and reliable tool. The FACT-G version 4 were utilized in many clinical trials as it is easy to complete and demonstrates sensitivity to the performance status and the extent of disease. Respondent rates the 27 items on the scale where each item is rated from (0) not at all to (4) very much. The scores of physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), and functional well-being (7 items) subscales range of 0-28, 0-28, 0-24, and 0-28, respectively. The highest score of that could be obtained on FACT-G is 108 where the highest the scores the better the quality of life of the patient. For the use in the current trail author obtain the LICENSING AGREEMENT from the copy-write owner.

Manipulation check: After each writing session, participants will be asked specific questions pertinent to how personal they feel their essays are and the degree to which they feel they have expressed their deep emotions in the writings. Each of these questions was rated on a 7-point scale.

Primary endpoint - The difference in the mean scores change of FACT-G from baseline to the end of second month between the two arms.

Secondary endpoint

- The difference in the mean scores change of FACT-G from baseline to the end of the second month within each arm.

Procedure, recruitment, and consent The recruitment will start in August 2021 and end in August 2024. Radiation and Medical Oncologists, breast surgeons and unite clark at Cancer center and SQUH will be briefed about the trail for they help in referring eligible patients to the trail. Participants who will be interested in participation will be contacted by the trial coordinator who will explain the study and screen potential participants for eligibility on the phone. Written informed consent will eventually obtained from all study participants. Participants will complete a baseline assessment that covers data related to clinical and socio-demographics , Medical and Surgical history and FACT-G. Given that participants come from different regions in Oman and to increase the feasibility of the intervention, assessments and experimental procedures will be performed via telephone in case participant could not be seen in person. For the intervention part, a "writing package" will be handed /emailed to every participant including blank paper with their identification numbers to be used for the writing task according to their assignment. Once participant done writing, they will scan and email back their writing to trail email address. After completing Assessment 1, participant will be scheduled for 3 writing consecutive days on which she will complete the writing task. In case participant is unable to schedule 3 consecutive days, 3 days will be scheduled proximally to each other within the same 1-week duration.

The process for the writing manipulation will as follows. On Day 1, a member of trail team will call the participant at a designated time and give a brief introduction to the writing task. Participant will be instructed to go to a quiet place in their house where no interruptions is expected. Then, participants will receive detailed standardized sets of instructions (as detailed below) based on existing work of Pennebaker. Thereafter, participant will be informed to start writing immediately after hanging up the phone and to write continuously for 20 min. The trail member will phone once 20 min lapsed. When writing session ends, the study member will call the participants to ask whether they experience any interruptions during the writing time. In case participant faces more than 5 min, she will be directed to continue writing till completing the 20-min writing time. Once finished, the participant will be asked to scan the writing paper and email it to trail email. Participant will be debriefed at the end by asking if she has any question or concerns. Then the writing time for the following day will be agreed upon. The above process will be repeated the second and third writing sessions, except for the initial introduction given on day 1. Outcome assessment with FACT-G will be conducted one and two months after finishing 3 writing sessions. After finishing the study, all participants will be debriefed. To maintain rapport with the participants and increase adherence to trial protocol, the same trail member will perform baseline assessments and give writing instructions for the same participant. Outcome assessment with FACT-G will be conducted one and two months after finishing 3 writing sessions by a blind assessor.

ELIGIBILITY:
Inclusion Criteria:

* Omani Women Having a breast cancer diagnosis stage, I and II
* Completing breast cancer surgery within 5 years
* Subsequently received adjuvant treatment including chemotherapy, hormonal treatment, or Radiation therapy
* Being comfortable writing and speaking in Arabic Or English

Exclusion Criteria:

* Nonconsenting
* Presence of severe physical illness
* Diagnoses with severe Mental or intellectual disorder
* Advanced breast cancer
* Un able to comply with trial protocol
* Presence of another cancer diagnoses

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The difference in the mean scores of Functional Assessment of Cancer Therapy general scale: FACT-G V4 | 1-3 MONTHS
  This 27-item measure examines the perceived quality of life across four dimensions including physical, social, emotional, and functional well-being in the past week. Each item is rated from (0) not at all to (4) very much. The scores of physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), and functional well-being (7 items) subscales range of 0-28, 0-28, 0-24, and 0-28, respectively. The highest score of that could be obtained on FACT-G is 108 where the highest the scores the better the quality of life of the patient

IPD SHARING:
Plan to Share IPD: Undecided